CLINICAL TRIAL: NCT03261414
Title: Prospective Randomized Study Evaluating the Effect of Pre-operative Hypnosis on Anesthesia, Analgesia and Perioperative Stress Laparoscopic Ileo-caecal Resections of Crohn's Disease.
Brief Title: HYSTERIA Evaluation of Clinical HYpnosis After Surgical Resection for Crohn Disease on Post-operative Analgesia
Acronym: HYSTERIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013_54; 2014-A00622-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-07-31; First posted 2017-08-25 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Inflammatory Bowel Diseases; Anesthesia
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With preoperative hypnosis (Experimental): standard care plus hypnosis followed by administration of propofol for anesthesia induction
  Interventions: Procedure: Hypnosis
- Without preoperative hypnosis (Active Comparator): standard care without preoperative hypnosis followed by administration of propofol for anesthesia induction
  Interventions: Procedure: usual care

INTERVENTIONS:
Procedure: Hypnosis — A short preanesthetic hypnosis before induction of anesthesia
  Arms: With preoperative hypnosis
Procedure: usual care — Standard care before induction of anesthesia
  Arms: Without preoperative hypnosis

SUMMARY:
The aim of this study will be to show a decrease in postoperative morphine consumption by the practice of perioperative self-hypnosis in patients undergoing laparoscopic ileo-caecal resection for Crohn's disease

ELIGIBILITY:
Inclusion Criteria:

* Being affected by a crohn's disease, reaching the small intestine (ileal or ileo-colic) and requiring ileo-caecal resection by laparoscopy
* Never been operated for abdominal crohn's disease

Exclusion Criteria:

* Pregnant women
* A history of intestinal resection for crohn's disease
* Emergency surgery
* Corticotherapy in progress
* Deaf patients
* non-Francophone Patients
* Patients with knowledge of self-hypnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | During the first 24 postoperative hours
  Compare the cumulative morphine consumption during 24 hours postoperative Data from PCA pump and patient medical record

SECONDARY OUTCOMES:
Total morphine consumption | between the 24 and the 48 postoperative hours
  Compare the cumulative morphine consumption between the 24 and the 48 postoperative hours Data from PCA pump and patient medical record
Total number of patients with complications | during first 7 postoperative days
Intraoperative consumption of hypnotics and opioids | during first 7 postoperative days
  The hypnotics and opioids drug dose will be recorded
Antiemetics consumption | during first 7 postoperative days
  The antiemetic drug dose will be recorded
Postoperative nausea and vomiting (PONV) Score | first 24 postoperative hours
  PONV risk assessment tool Based on apfel's simplified risk score
Duration of hospital stay | during first 7 postoperative days
Time physiological function recovery | during first 7 postoperative days
  Ability to drink, to eat, to urinate, to walk

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Zerbib, MD,PhD, Principal Investigator — University Hospital of Lille
Locations (1):
- Hôpital Claude Huriez, Lille, France

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391